CLINICAL TRIAL: NCT03795636
Title: Allium Sativum Extract as an Irrigant in Pulpectomy of Primary Molars: 12 Month In-vivo Study
Brief Title: Allium Sativum Extract as an Irrigant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmad Elheeny, Lecturer of pediatric dentistry, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 307
Record Dates: First submitted 2019-01-02; First posted 2019-01-08 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Infected Root Canals of Primary Molars
Keywords: Primary molars; Garlic extract; Sodium hypochlorite; Pulpectomy
MeSH Terms: interventions — PMK-S005

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Device: No

ARMS (2):
- Garlic extracts root canal irrigation group (Experimental): Experimental group treated with garlic extract
  A 100 gram of garlic cloves has been cleaned, peeled and dried. Ethanol of 70% concentration was added for 60 seconds. The cloves were placed in a laminar airflow chamber for evaporation of residual ethanol. Using a sterile mortar and pestle, cloves were homogenized aseptically and filtered through a double layer paper. The fully concentrated extracted was diluted to the concentration of 25% with distilled water
  Interventions: Other: Garlic extract
- Sodium hypochlorite root canal irrigation group (Active Comparator): Control group which treated conventionally using .5 ml of 5.25% NaOCl (COLTENE®ENDO, Switzerland)
  Interventions: Other: NaOCl (COLTENE®)

INTERVENTIONS:
Other: Garlic extract — A 100 gram of garlic cloves has been cleaned, peeled and dried. Ethanol of 70% concentration was added for 60 seconds. The cloves were placed in a laminar airflow chamber for evaporation of residual ethanol. Using a sterile mortar and pestle, cloves were homogenized aseptically and filtered through a double layer paper. The fully concentrated extracted was diluted to the concentration of 25% with distilled water
  Arms: Garlic extracts root canal irrigation group
Other: NaOCl (COLTENE®) — Sodium hypochlorite
  Arms: Sodium hypochlorite root canal irrigation group

SUMMARY:
Garlic extract as herbal compound has potent antibacterial properties and can be used safely as an irrigant for pulpectomy procedure of primary molars root canals with high clinical and radiographic outcomes

DETAILED DESCRIPTION:
Aim: This study indented to assess the clinical and radiographic assessment of garlic extract as an intracanal irrigant for pulpectomy of primary molars.

Methodology: 91 child with 100 teeth submitted into this study were equally categorized into the test group (group 1) which irrigated with garlic extract and control group (group 2) that received sodium hypochlorite (NaOCl). Then, each group has been subjected to further specification according to the tooth preoperative clinical and radiographic features into has been into 2 subgroups. Clinical and radiographic success rates were checked at 3, 6 and 12 months. Fisher's exact test for binary variable was used for data analysis with p-value ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Class I or II according to American Society of Anesthesiologists (ASA)
2. Irreversible pulpititis recognised through; (1) profuse bleeding from root canal orifices after complete debridement of coronal pulp tissue and cannot be dominated by moist cotton pellet. (2) History of lingered thermal pain spontaneous nocturnal pain
3. Necrotic pulp tissues which may be asymptomatic or manifested with dull ache pain
4. Pathological tooth mobility
5. Percussion sensitivity
6. Swelling close to involved tooth accompanied with or without fistula Radiographic characteristics of the root and supporting structures

1. Normal radiographic findings

2. Interruption of lamina dura

3. Furcation radiolucency

Exclusion Criteria:

* Specifications of exclusion

  1. Uncooperativeness of child and/or parents or caregivers behavior
  2. Unrestorable tooth
  3. Presence of internal root resorption
  4. Presence of calcific metamorphosis inside root canals
  5. Presence of root resorption exceeding one third of its length

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2016-10-30 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
oral examination | 12 months
  Pain assessment using Visual Analog Score for pain
radiographic success or failure | 12 months
  Radiographic assessment using periapical radiograph and score (0) applied for absence of radiolucency and score (1) for presence of radiolucency

SECONDARY OUTCOMES:
Types of failures | 12 months
  detecting the percent of different failure types accompanied with pulpectomy procedures after using garlic as an irrigant solution.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elheeny AAH. Allium sativum extract as an irrigant in pulpectomy of primary molars: A 12-month short-term evaluation. Clin Exp Dent Res. 2019 Jun 26;5(4):420-426. doi: 10.1002/cre2.197. eCollection 2019 Aug. PMID 31452953